CLINICAL TRIAL: NCT06576908
Title: Evaluation of Image Quality From an On-Couch, Cone Beam Computed Tomography (CBCT) Radiation Treatment System for Image Guidance and Treatment Adaptation
Brief Title: Evaluation of On-Couch CBCT Image Quality
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Varian, a Siemens Healthineers Company (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: VAR-2023-07
Record Dates: First submitted 2024-07-26; First posted 2024-08-29 (Actual); Last update posted 2024-12-03 (Actual); Status verified 2024-11

CONDITIONS: Head and Neck Cancer; Thoracic Cancer; Abdominal Cancer; Pelvic Cancer
MeSH Terms: conditions — Head and Neck Neoplasms; Pelvic Neoplasms

STUDY DESIGN:
Intervention Model Description: This is a prospective, single-arm, single-site study designed to generate data describing the image quality and applicability/useability of a high-performance, on-couch CBCT imaging technology in patients receiving radiation treatment for cancer.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (1):
- HyperSight Imaging arm (Experimental): Subjects have both HyperSight and conventional CBCT imaging.
  Interventions: Device: HyperSight Imaging

INTERVENTIONS:
Device: HyperSight Imaging — Subjects receive both HyperSight imaging and conventional imaging, on their first day of radiation treatment, on their second day of treatment, and on their last day of treatment.

SUMMARY:
This is a prospective, single-arm, single-site study designed to generate data describing the image quality and applicability/useability of a high-performance, on-couch CBCT imaging technology (HyperSight) in patients receiving radiation treatment for cancer on a C-arm linear accelerator (TrueBeam).

ELIGIBILITY:
Inclusion Criteria:

* Patient age is ≥ 18 years old.
* Patient has a diagnosis of primary or metastatic cancer, including but not limited to tumors arising from or involving the head/neck, lungs, liver, pancreas, prostate, urinary bladder, rectum, cervix or uterus.
* A previous (standard-of-care) decision was made to treat the patient with radiation therapy using a Varian TrueBeam treatment system.
* A previous (standard-of-care) decision was made to treat the patient with a radiation dose of at least 20 Gy in at least 5 fractions, one fraction per day on consecutive days, Monday to Friday.
* Patient is willing and able to provide informed consent to participate in the study.

Exclusion Criteria:

* Patient is pregnant or has plans for pregnancy during the period of treatment.
* Patient is part of a vulnerable population (per ISO 14155:2020, "individuals who are unable to fully understand all aspects of the investigation that are relevant to the decision to participate, or who could be manipulated or unduly influenced as a result of a compromised position, expectation of benefits or fear of retaliatory response").

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 46 (Estimated)
Dates: Start 2024-10-17 (Actual); Primary Completion 2025-10 (Estimated); Study Completion 2025-12 (Estimated)

PRIMARY OUTCOMES:
Comparison of overall free-breathing image quality: HyperSight CBCT vs Conventional CBCT | Day 1 of radiation treatment, day 2 of radiation treatment, and the last day of radiation treatment (up to 6 weeks after the start of treatment).
  Semi-quantitative scoring (5-point Likert scale) of on-treatment, free-breathing HyperSight-TrueBeam CBCT images compared to on-treatment, free-breathing conventional TrueBeam CBCT images by three independent observers. The Likert scale values will represent a range of opinion from strong preference for HyperSight-TrueBeam CBCT images to strong preference for conventional TrueBeam CBCT images.

SECONDARY OUTCOMES:
Comparison of overall image quality: HyperSight CBCT vs Computed Tomography (CT) simulation images | Day 1 of radiation treatment, day 2 of radiation treatment, and the last day of radiation treatment (up to 6 weeks after the start of treatment).
  Semi-quantitative scoring (5-point Likert scale) of on-treatment HyperSight-TrueBeam CBCT images compared to pre-treatment, diagnostic-quality, planning CT images by three independent observers. The Likert scale values will represent a range of opinion from strong preference for HyperSight-TrueBeam CBCT images to strong preference for planning CT images.
Comparison of motion artifacts: HyperSight CBCT vs. Conventional CBCT | Day 1 of radiation treatment, day 2 of radiation treatment, and the last day of radiation treatment (up to 6 weeks after the start of treatment).
  Semi-quantitative scoring (5-point Likert scale) of motion artifacts in HyperSight-TrueBeam CBCT images compared to on-treatment conventional TrueBeam CBCT images by three independent observers. The Likert scale values will represent a range of opinion from strong preference for HyperSight-TrueBeam CBCT images to strong preference for conventional TrueBeam CBCT images.
Comparison of metal artifacts: HyperSight CBCT vs. Conventional CBCT | Day 1 of radiation treatment, day 2 of radiation treatment, and the last day of radiation treatment (up to 6 weeks after the start of treatment).
  Semi-quantitative scoring (5-point Likert scale) of metal artifacts in HyperSight-TrueBeam CBCT images compared to on-treatment conventional TrueBeam CBCT images by three independent observers. The Likert scale values will represent a range of opinion from strong preference for HyperSight-TrueBeam CBCT images to strong preference for conventional TrueBeam CBCT images.
Comparison of overall breath hold image quality: HyperSight CBCT vs Conventional CBCT | Day 1 of radiation treatment, day 2 of radiation treatment, and the last day of radiation treatment (up to 6 weeks after the start of treatment).
  Semi-quantitative scoring (5-point Likert scale) of on-treatment, breath-hold HyperSight-TrueBeam CBCT images compared to on-treatment, breath-hold conventional TrueBeam CBCT images by three independent observers. The Likert scale values will represent a range of opinion from strong preference for HyperSight-TrueBeam CBCT images to strong preference for conventional TrueBeam CBCT images.
Comparison of Hounsfield Unit accuracy: HyperSight CBCT vs Conventional CBCT and CT Simulation images | Day 1 of radiation treatment, day 2 of radiation treatment, and the last day of radiation treatment (up to 6 weeks after the start of treatment).
  The HU accuracy of clinical HyperSight-TrueBeam CBCTs will be evaluated by comparing mean HUs and SDs for regions of interest in different tissue types (muscle, fat, lungs, and bones) on the planning CTs, HyperSight-TrueBeam CBCTs, and conventional TrueBeam CBCT.
Patient's perspectives of on-treatment HyperSight-TrueBeam CBCT | Day 1 of radiation treatment and the last day of radiation treatment (up to 6 weeks after the start of treatment).
  Semi-structured interview integrating the validated six-item State Anxiety scale derived from the State-Tait Anxiety Inventory.
Patient tolerability of on-treatment, breath-hold HyperSight-TrueBeam CBCT imaging. | Day 1 of radiation treatment, day 2 of radiation treatment, and the last day of radiation treatment (up to 6 weeks after the start of treatment).
  Proportion of patients able to complete HyperSight-TrueBeam CBCT breath-hold imaging in a single breath-hold compared to conventional TrueBeam CBCT breath-hold imaging.
Patient tolerability of on-treatment, breath-hold HyperSight-TrueBeam CBCT imaging. | Day 1 of radiation treatment, day 2 of radiation treatment, and the last day of radiation treatment (up to 6 weeks after the start of treatment).
  Number of breath-holds required to complete HyperSight-TrueBeam CBCT breath-hold imaging compared to conventional TrueBeam CBCT breath-hold imaging.
Breath hold imaging time | Day 1 of radiation treatment, day 2 of radiation treatment, and the last day of radiation treatment (up to 6 weeks after the start of treatment).
  Total HyperSight-TrueBeam CBCT breath-hold image acquisition time compared to conventional TrueBeam CBCT breath-hold imaging.

CONTACTS AND LOCATIONS:
Locations (1):
- Princess Margaret Cancer Centre (University Health Network), Toronto, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No